CLINICAL TRIAL: NCT05665608
Title: Prevention Of Sudden Cardiac Death After Myocardial Infarction by Defibrillator Implantation
Acronym: PROFID EHRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Daniela Fischer, Project Manager, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHS-2019-0209
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sudden Cardiac Death; Myocardial Infarction
Keywords: Implantable Cardioverter Defibrillator; Sudden Cardiac Death; Myocardial Infarction
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Infarction | interventions — Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: An investigator-driven, prospective, parallel-group, randomised, open, blinded outcome assessment (PROBE), multi-centre, non-inferiority trial without investigational medical products (Proof of Strategy Trial)
Masking Description: The PROFID EHRA trial is an open-label, blinded outcome assessment study. Thus, unblinding procedures for investigators are not applicable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Therapy with ICD device therapy (Active Comparator): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure / chronic coronary syndromes and will receive an ICD device
  Interventions: Device: Implantable cardioverter-defibrillator (ICD); Drug: Optimal Medical Therapy (OMT)
- Optimal Medical Therapy without ICD device therapy (Experimental): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure / chronic coronary syndromes and will not receive an ICD device
  Interventions: Drug: Optimal Medical Therapy (OMT)

INTERVENTIONS:
Device: Implantable cardioverter-defibrillator (ICD) — A transvenous ICD consists of an electronic medical device and electrode leads. Besides the possibility to shock during arrhythmias the ICD can potentially terminate ventricular tachycardias by rapid pacing for short periods (small bursts of pacing).
  The subcutaneous defibrillator is an established and valid alternative to the transvenous ICD for the prevention of SCD, but in patients without an indication for bradycardia support, cardiac resynchronisation or antitachycardia pacing.
  The extravascular implantable cardioverter-defibrillator (EV ICD) system with substernal lead placement is a novel nontransvenous alternative to current available transvenous and subcutaneous ICDs.
  Arms: Optimal Medical Therapy with ICD device therapy
Drug: Optimal Medical Therapy (OMT) — Patients will be treated according to Optimal Medical Therapy defined by the following guidelines:
  1. 2019 ESC guidelines for the diagnosis and management of chronic coronary syndromes
  2. 2021 ESC guidelines for the diagnosis and treatment of acute and chronic heart failure

SUMMARY:
Patients who have survived a myocardial infarction (MI) are at increased risk for sudden cardiac death (SCD) caused by ventricular tachycardia and ventricular fibrillation. A severely reduced left ventricular ejection fraction (LVEF) as a rough overall measure of impaired heart function after MI was shown to indicate a higher risk for SCD. Based on this observation, two landmark randomised trials, MADIT II and SCD-HeFT, were conducted between end of the 1990s and early 2000s. These trials compared the survival of patients with severely reduced LVEF who received an implantable cardioverter-defibrillator with the survival of patients being on medical therapy alone. They reported a significantly better survival of patients in the defibrillator arm and led to international guideline recommendations for routine implantation of defibrillators in survivors of MI with severely impaired LVEF as a means for primary prevention of SCD. Since then, the management of these patients has changed dramatically with the advent of a series of novel drug classes that reduce not only mortality but specifically SCD leading to a substantial decrease of the sudden death rates as well as of the rates of appropriate defibrillator therapies implanted for primary prevention of SCD. At the same time, the complication rates associated with the defibrilllator therapy remain significant without obvious decrease. Thus, the risk-benefit of routine defibrillator implantation for primary prevention of SCD in patients with severely reduced LVEF has substantially changed since the conduction of the landmark trials that established this therapy. Due to the inherent risks and considerable costs of the defibrillator, a novel randomised adequately powered assessment of the potential benefit or harm of the defibrillator in survivors of MI with reduced LVEF under contemporary optimal medical treatment (OMT) appears imperative.

OBJECTIVE:

To demonstrate that in post-MI patients with symptomatic heart failure who receive OMT for this condition, and with reduced LVEF ≤ 35%, OMT without ICD implantation (index group) is not inferior to OMT with ICD implantation (control group) with respect to all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Naïve to implantation of any pacemaker or defibrillator
3. Documented history of MI either as ST segment elevation myocardial infarction (STEMI) or as non-ST segment elevation myocardial infarction (NSTEMI) at least 3 months prior to enrolment.
4. Symptomatic heart failure with New York Heart Association (NYHA) class II or III.
5. On OMT for at least 3 months prior to enrolment.
6. LVEF ≤ 35% (at transthoracic echocardiography or cardiac magnetic resonance imaging [MRI] at least 3 months after MI).
7. Signed informed consent.

Inclusion criterion I3 defines myocardial infarction according to the 2018 ESC/ACC/AHA/WHF Fourth Universal Definition of myocardial infarction

Exclusion Criteria:

1. Class I or IIa indication for implantation of an ICD for secondary prevention of SCD and ventricular tachycardia.
2. Ventricular tachycardia induced in an electrophysiologic study.
3. Unexplained syncope when ventricular arrhythmia is suspected as the cause of syncope.
4. Class I or IIa indication for Cardiac Resynchronization Therapy (CRT)
5. Foreseable violation of instruction for use (IFU) of the ICD device selected for implantation (valid for control group patients, only).
6. Acute coronary syndrome or coronary angioplasty or coronary artery bypass grafting performed within 6 weeks prior to enrolment.
7. Cardiac valve surgery or percutaneous cardiac valvular intervention performed within 6 weeks prior to enrolment.
8. On the waiting list for heart transplantation.

   Class I or IIa indication for implantation of an ICD for secondary prevention of SCD and ventricular tachy-cardia has to be assessed according to the 2022 ESC Guidelines for the management of patients with ven-tricular arrhythmias and the prevention of SCD.
9. Any known disease that limits life expectancy to less than 1 year.
10. Participation in another randomised clinical trial if study-specific treatment is still active at enrolment into PROFID EHRA.
11. Previous participation in PROFID EHRA.

Parallel participation in sub-studies connected to this trial is permitted as well as in purely observational studies without any pre-defined intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3595 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Time from randomisation to the occurrence of all-cause death. | event-driven, expected about 15 months after last patient in
  Randomization to end of study

SECONDARY OUTCOMES:
Time from randomisation to death from cardiovascular causes | Randomization to end of study (event-driven, expected about 15 months after last patient in
  Time from randomisation to death from cardiovascular causes
Time from randomisation to sudden cardiac death | Randomization to end of study (event-driven, expected about 15 months after last patient in
  Time from randomisation to sudden cardiac death
Time from randomisation to first hospital readmissions for cardiovascular causes after date of randomisation | Randomization to end of study (event-driven, expected about 15 months after last patient in
  Time from randomisation to first hospital readmissions for cardiovascular causes after date of randomisation
Average length of stay in hospital during the study period | Randomization to end of study (event-driven, expected about 15 months after last patient in
  Average length of stay in hospital during the study period
Quality of life (EQ-5D-5L) trajectories over time | At baseline and 12-month intervals thereafter
  Quality of life (EQ-5D-5L) trajectories over time

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof, Principal Investigator — Deutsches Herzzentrum der Charité, Department of Cardiology, Angiology and Intensive Care Medicine; Nikolaos Dagres, MD, Principal Investigator — Deutsches Herzzentrum der Charité, Department of Cardiology, Angiology and Intensive Care Medicine
Locations (86):
- Austria (9):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - LKH Universitätsklinikum Graz, Graz
  - Tirol Kliniken - Universitätsklinik Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Landeskrankenhaus Salzburg - Universitätsklinikum der PMU, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - Universitätsklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (4):
  - OLV Ziekenhuis Campus Aalst, Aalst
  - AZ Sint-Jan Brugge-Campus Sint-Jan, Bruges
  - Centre hospitaliser régional (CHR) de la Citadelle, Liège
  - Centre Hospitalier Universitaire CHU UCL Namur - Site Godinne, Yvoir
- Czechia (4):
  - Fakultní Nemocnice Olomouc, Olomouc
  - Všeobecná Fakultní Nemocnice v Praze, Prague
  - Institut Klinické a Experimentální Medicíny, Prague
  - Masaryk Hospital, Ústí nad Labem
- Aarhus University Hospital I, Aarhus, Denmark
- France (10):
  - CHU Amiens Picardie, Amiens
  - Hôpital de la Cavale Blanche-CHU BREST, Brest
  - CHU Henri Mondor, Créteil
  - University Hospital Grenoble-Alpes, Grenoble
  - Européen Georges Pompidou Hospital Paris, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Chu de Rennes, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - University Hospital Rangueil Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (37):
  - St. Marien-Krankenhaus - Klinikum Westmünsterland, Ahaus
  - Helios Klinikum Aue, Aue
  - Kerckhoff-Klinik Bad Nauheim, Bad Nauheim
  - Herz- und Diabeteszentrum NRW Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Segeberger Kliniken Gmbh, Bad Segeberg
  - Charité - Universitätsmedizin Berlin (CCM), Berlin
  - Sana Klinikum Lichtenberg, Berlin
  - Charité - Universitätsmedizin Berlin (CBF), Berlin
  - BG Klinikum Unfallkrankenhaus Berlin, Berlin
  - Charité - Universitätsmedizin Berlin (CVK), Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Klinikum Bielefeld, Bielefeld
  - REGIOMED Klinikum Coburg, Coburg
  - Carl-Thiem-Klinikum, Cottbus
  - Städtisches Klinikum Dresden, Dresden
  - Technische Universität Dresden - Herzzentrum Dresden, Dresden
  - Elisabeth-Krankenhaus Essen, Essen
  - Georg-August-Universität Göttingen - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Klinikum Gütersloh, Gütersloh
  - Asklepios Kliniken Hamburg, Hamburg
  - Asklepios Klinikum Harburg, Hamburg
  - Albertinen Herz- und Gefäßzentrum, Hamburg
  - Universitätsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - B.Braun Ambulantes Herzzentrum Kassel, Kassel
  - Asklepios Kliniken Langen, Langen
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum St. Georg, Leipzig
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Johannes Wesling Klinikum, Minden
  - Klinikum der Ludwig-Maximilians-Universität München (LMU Klinikum), München
  - FEK - Friedrich-Ebert-Krankenhaus Neumünster, Neumünster
  - Klinik Rothenburg ANregiomed, Rothenburg upon Tauber
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Semmelweis University, Budapest, Hungary
- Rambam Health Care Campus, Haifa, Israel
- Le Centre Hospitalier Universitaire de Martinique, Fort-de-France Cedex, Martinique
- Netherlands (5):
  - Amsterdam UMC, Amsterdam
  - Stichting Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
- Poland (3):
  - Kliniczny Szpital Wojewódzki Nr 2 im.Św.Jadwigi Królowej w Rzeszowie, Rzeszów
  - Wojskowy Instytut Medyczny, Warsaw
  - Śląskie Centrum Chorób Serca w Zabrzu, Zabrze
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante
  - Instituto de Investigación Hospital 12 de Octubre, Madrid
  - La Paz University Hospital, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
- United Kingdom (6):
  - Calderdale Royal Hospital, Halifax
  - The Leeds Teaching Hospitals NHS Trust - St James's University Hospital, Leeds
  - Queen Elizabeth The Queen Mother Hospital Margate, Margate
  - George Eliot Hospital, Nuneaton
  - Salisbury District Hospital, Salisbury
  - University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qian Y, Roque CR, Woods B, Iglesias Urrutia CP, Gc VS, Gur Arie M, Fischer D, Dagres N, Hindricks G, Manca A. Economic evaluation protocol for the PRevention Of sudden cardiac death aFter myocardial Infarction by Defibrillator implantation: the PROFID EHRA trial. BMJ Open. 2026 Jan 8;16(1):e097495. doi: 10.1136/bmjopen-2024-097495. PMID 41506764
- [Derived] Dagres N, Gale CP, Nadarajah R, Boveda S, Merino JL, Nielsen JC, Kirchhof P, Kutyifa V, Taborsky M, Thiele H, Tijssen JGP, Verma A, De Potter T, Braunschweig F, Merkely B, Sommer P, Vernooy K, Suleiman M, Purerfellner H, Hindricks G; PROFID EHRA trial investigators. PRevention of sudden cardiac death aFter myocardial infarction by defibrillator implantation: Design and rationale of the PROFID EHRA randomized clinical trial. Am Heart J. 2026 Jan;291:37-43. doi: 10.1016/j.ahj.2025.07.071. Epub 2025 Aug 6. PMID 40774643